CLINICAL TRIAL: NCT04275219
Title: Safety and Efficacy of the Tong-Fu-Xing-Shen Herbal Formula for Stroke-Associated Pneumonia (TFXSHF)
Brief Title: Safety and Efficacy of the Tong-Fu-Xing-Shen Herbal Formula for Stroke-Associated Pneumonia
Acronym: TFXSHF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Collaborators: People's Hospital of Ganzhou City (Unknown); People's Hospital of Lianjiang City (Unknown); Yangjiang Hospital of Traditional Chinese Medicine (Unknown); Shenyang No. 2 Hospital of Traditional Chinese Medicine (Unknown); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 001/20180101
Record Dates: First submitted 2020-02-11; First posted 2020-02-19 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-05

CONDITIONS: Stroke; Complication
Keywords: stroke-associated pneumonia; Tong-Fu-Xing-Shen herbal formula; Traditional Chinese medicine; Brain-gut-lung axis; Randomized controlled trial
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tong-Fu-Xing-Shen herbal formula (Experimental): Tong-Fu-Xing-Shen herbal formula prescription (0.4g*36 capsules/bottle，1-4 capsules each time, three times a day.) for 10-12days.
  Interventions: Drug: Tongfu capsules
- The Placebo of Tong-Fu-Xing-Shen herbal formula (Placebo Comparator): The Placebo of Tong-Fu-Xing-Shen herbal formula prescription (0.4g*36 capsules/bottle，1-4 capsules each time, three times a day.) for 10-12 days.
  Interventions: Drug: The Placebo of Tongfu capsules

INTERVENTIONS:
Drug: Tongfu capsules — Tongfu capsules include 5 herbals
  Arms: Tong-Fu-Xing-Shen herbal formula
Drug: The Placebo of Tongfu capsules — The Placebo of Tongfu capsules are made from dextrin, starch and so on.
  Arms: The Placebo of Tong-Fu-Xing-Shen herbal formula

SUMMARY:
Stroke-associated pneumonia (SAP) is the major complication of acute intracerebral haemorrhage (AICH), leads to poor clinical outcomes and increases the financial burden on the medical system. Prophylactic antibiotics do not reduce the mortality rate of SAP. The Tong-Fu-Xing-Shen herbal formula (TFXS) was shown to be effective for the prevention and treatment SAP in a previous clinical trial. To clarify whether TFXS is effective and safe for the treatment of SAP and affects the immunological mechanism of the "brain-gut-lung" pathway of SAP, the investigators designed this study.

DETAILED DESCRIPTION:
This is a multicentre, randomized, double-blind, placebo-controlled clinical trial. A total of 218 patients will be recruited and randomly assigned to the experimental group (EG) or the control group (CG) in a 1:1 ratio. The treatment course will be 10-12 consecutive days, with a 90±7-day follow-up. The primary outcome is the all-cause mortality rate and the mortality of pneumonia at the 90±7-day follow-up. Secondary outcomes include changes in the gut microbiota; changes in the NIHSS score, BI index, mRS score, and Stroke-Specific Quality of Life scale (SS-QOL) score; and so on.

ELIGIBILITY:
Inclusion criteria

For inclusion, participants will need to fulfil all the following criteria:

1. A diagnosis of intracerebral haemorrhage according to 2019 Chinese guidelines for the diagnosis and treatment of acute intracerebral haemorrhage [9], with a CT scan of the brain confirming acute intracerebral haemorrhage;
2. Age between 18 and 85;
3. A diagnosis of SAP according to the modified CDC standard [10];
4. Within 7 days after stroke onset; and
5. Willingness to participate and to sign the informed consent form.

Exclusion criteria

Participants with any of the following conditions will be excluded:

1. Cerebral haemorrhage is confirmed by examination to be caused by a brain tumour, brain trauma, blood disease, cerebrovascular malformation (a congenital abnormality) or aneurysm;
2. Cerebral herniation;
3. A GCS score <7;
4. Any antibiotic treatment within 4 weeks before the start of the study;
5. Pulmonary tuberculosis, pulmonary oedema, pulmonary embolism, noninfectious pulmonary oedema or respiratory circulation failure;
6. Liver or kidney function parameters (such as alanine aminotransferase [ALT], aspartate aminotransferase [AST] and creatinine [Cre]) 3 times higher than the upper limit of normal;
7. A clear history of gastrointestinal diseases, such as gastrointestinal tumours and inflammatory bowel disease, or a gastrointestinal bleeding period within 3 months;
8. Immune-related diseases, such as SLE, rheumatoid arthritis, and Sjogren's syndrome, or receiving immunotherapy for other diseases; and
9. Unsuitable for the trial as decided by the researchers.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Estimated)
Dates: Start 2019-03-15 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
the all-cause mortality rate | 90±7 days
  Any cause of death
the mortality of stroke associated pneumonia | 90±7 days
  the death of stroke associated pneumonia

SECONDARY OUTCOMES:
changes in the gut microbiota between the experiment group and the control group | Baseline (before drug), after drug 10-12 days
  gut microbiota is monitored via 16S rRNA gene sequence analysis
National Institute of Health of stroke scale （NIHSS） | Baseline (before drug), after drug 10-12 days, 90±7 days
  The NIHSS is for evaluation of neurological deficits. The NIHSS includes the following domains: level of conscious-ness, eye movements, integrity of visual fields, facial movements,arm and leg muscle strength, sensation, coordination, language,speech and neglect. Each impairment is scored on an ordinal scaleranging from 0 to 2, 0 to 3, or 0 to 4. The scoing of it ranges from 0 to 42. The higher scoring represents the more serious nerve defects. The scoring from 0-1 are normal or close to normal, 2-4 are mild, 5-15 are moderate, 6-20 are medium and severe and more than 20 points are severe neurological dysfunction.
Stroke Specific Quality Of Life scale (SS-QOL) (SS-QOL) score | 90±7 days
  The Stroke Specific Quality Of Life scale (SS-QOL) is a patient-centered outcome measure intended to provide an assessment of health-related quality of life (HRQOL) specific to patients with stroke.It consists of 49 items in the 12 domains of energy, family roles, language, mobility, mood, personality, self-care, social roles, thinking, upper extremity (UE) function, vision, and work/productivity.
  The score ranges from 0 to 100. The higher the score, the better the quality of life.
Barthel index | Baseline (before drug), after drug 10-12 days, 90±7 days
  The score ranges from 0 to 100. It represents the self-care ability. BI index ≤40 defines heavily dependent, ranges from 41 to 60 defines moderate dependent, ranges from 61 to 99 defines mild dependent and 100 defines independent. The scoring ≥<90 defines life cannot be independent. The percentage of BI 100-90 points in the three groups was statistically followed up by 90ds. The higher scoring represents a better outcome. There are 4 evaluation grades for 10 aspects(complete independence，part of the help, great help, absolutely dependent).The 10 aspects of the BI index includes eating(10,5,0,0), washing(5,0,0,0), making up（5,0,0,0）, dressing up(10,5,0,0），control of the stool(10,5,0,0), control of the urination(10,5,0,0), going to toilet(10,5,0,0), bed-chair transform(15,10,5,0), walking on the ground(15,10,5), going up and down the stairs(10,5,0,0).
Modified rankin scale (mRS) | after drug 10-12 days, 90±7 days
  It represents the recovery of neural functions. The scoring ranges from 0 to 5. Scoring 2-5 is defined as disability, which can be divided into 4 grades: mild, moderate, severe and severe.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Province Hospital of Tradtional Chinese Medicine, Guangzhou, Guangdong, China